CLINICAL TRIAL: NCT05488886
Title: Optimizing the Bioavailability and Metabolism of Aronia Berry Polyphenols for Improving Gut Health
Brief Title: Bioavailability of Aronia Berry Polyphenols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-0702; Protocol Version 07/01/2022 (Other: UW Madison); A074000 (Other: UW Madison)
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Gut Health; Metabolism; Polyphenols

STUDY DESIGN:
Intervention Model Description: The order of intervention foods (A-D) will be randomized for each participant upon study enrollment. Wash-in and wash-out periods are 6 days long, and food consumption and sampling durations are 24 hours.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: Whole Aronia Berry Powder (Experimental)
  Interventions: Dietary Supplement: Whole Aronia Berry Powder Applesauce
- B: Aronia Berry Extract (Experimental)
  Interventions: Dietary Supplement: Aronia Berry Extract Applesauce
- C: Phospholipid-Polyphenol (Experimental)
  Interventions: Dietary Supplement: Phospholipid-Polyphenol Applesauce
- D: Low-Polyphenol Control (Experimental)
  Interventions: Other: Low-Polyphenol Control Applesauce

INTERVENTIONS:
Dietary Supplement: Whole Aronia Berry Powder Applesauce — The food will be designed to be a berry-flavored applesauce. The food will include applesauce, sweeteners, citric acid, natural flavors and food colorants. Applesauce A will additionally contain whole aronia berry powder (Milne MicroDried, Nampa, ID).
  Arms: A: Whole Aronia Berry Powder
Dietary Supplement: Aronia Berry Extract Applesauce — The food will be designed to be a berry-flavored applesauce. The food will include applesauce, sweeteners, citric acid, natural flavors and food colorants. Applesauce B will additionally contain aronia berry extract (Artemis International, Fort Wayne, IN).
  Arms: B: Aronia Berry Extract
Dietary Supplement: Phospholipid-Polyphenol Applesauce — The food will be designed to be a berry-flavored applesauce. The food will include applesauce, sweeteners, citric acid, natural flavors and food colorants. Applesauce C will additionally contain PLP which will be prepared with commercially-available aronia juice concentrate (Greenwood Associates, Niles, IL) and soy lecithin (Whole Foods, Austin, TX).
  Arms: C: Phospholipid-Polyphenol
Other: Low-Polyphenol Control Applesauce — The food will be designed to be a berry-flavored applesauce. The food will include applesauce, sweeteners, citric acid, natural flavors and food colorants. Applesauce D will not contain additional polyphenol-rich ingredients and is thus considered a low-polyphenol control.
  Arms: D: Low-Polyphenol Control

SUMMARY:
The objective of this study is to conduct a randomized cross-over dietary intervention among healthy adults to compare the bioavailability and the fecal polyphenol metabolites of intervention foods made with whole aronia berry powder, aronia berry extract, phospholipid-polyphenol (PLP), and a low-polyphenol control. 10 participants will be enrolled and can expect to be on study for up to 28 days.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD): Crohn's disease and ulcerative colitis are two conditions of IBD that are characterized by chronic inflammation and damage of the gastrointestinal tract. In the United States alone, IBD are estimated to affect as many as 1.6 million people. IBD are associated with high morbidity, decreased quality of life, as well as substantial health care costs. IBD currently have no known cure, and treatment of IBD often requires the use of potent immunosuppressors which may lead to side effects or surgery.

Berries and prevention of chronic inflammation: Anthocyanins and other polyphenols are promising dietary agents to prevent and treat IBD by improving intestinal barrier dysfunction, inhibiting differentiation of pro-inflammatory T cells, reducing production of proinflammatory cytokines, and preventing oxidative stress. While preliminary studies are promising, translational human intervention studies are needed to refine delivery of polyphenol-rich foods and to confirm anti-inflammatory mechanisms.

Berries are rich dietary sources of polyphenols and essential nutrients. Polyphenol intake varies significantly by dietary patterns, but mean intake is estimated ~900 mg/day. Among berries, the polyphenol-dense aronia berry is one of the richest sources of fruit polyphenols.

Challenges associated with aronia berry consumption: In spite of its beneficial nutritional properties, the consumption of large amounts of whole aronia berry is not practical because of significant sorbitol and fiber content, which could lead to gastrointestinal discomfort for some individuals. Particularly, IBD patients often are required to limit fiber and whole fruit intake. The investigator's research group recently developed a novel method to extract polyphenols from fruit juice using food-grade lecithin which overcomes this problem.

The investigators hypothesize the resulting phospholipid-polyphenol (PLP) enriched material can improve the delivery of anthocyanins to the gut relative to a purified extract, and similar to that of whole berry. The aim of this study is to determine the comparative metabolism and bioavailability of aronia berry PLP intervention to extract, whole berry, and control food.

Consumption of Intervention Foods: In the morning of the day of each intervention and sampling period (days 6, 13, 20, and 27 i), participants will be asked to visit the Bolling Laboratory at the Department of Food Science fasted. Participants will then be asked to empty their bladders and then consume one serving of the applesauce (≤200 g). Then, in the next 24 h, participants will be asked to only consume commercially available frozen and shelf-stable low-polyphenol meals and snacks provided by study personnel. Insulated bags will be provided to participants for transport of frozen meals. The low-polyphenol diet and snacks will consist of dairy products, meat, low-phenolic snacks (e.g., banana, potato chips) and starch sources (e.g. white bread, rice, and plain bagels). Water will be available to participants over the time course, and its intake is not restricted.

ELIGIBILITY:
Inclusion Criteria:

* willing to consume low-anthocyanin diets during the last days of wash-in and wash-out periods
* willing to consume intervention foods during the sampling periods
* willing to provide 24-hour urine and fecal samples during the sampling periods.

Exclusion Criteria:

* people who do not consider themselves healthy
* anyone with a self-reported previous diagnosis of a gastrointestinal disease (e.g. inflammatory bowel disease, irritable bowel syndrome)
* undergoing current cancer treatment (i.e., chemotherapy, radiation therapy)
* are pregnant, lactating, or trying to become pregnant
* unwilling to consume study foods, or are allergic to sunflower, food colorants, berry ingredients, or any other component of the study foods.
* taking medication that contraindicates grapefruit juice consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Urinary Polyphenol Catabolite Concentration | sampled on day 6, 13, 20, and 27 (participant randomized to different interventions each visit)
  Targeted analysis of free urinary polyphenol metabolites will be performed by ultra-high performance liquid chromatography tandem mass spectrometry (UHPLC-MS/MS).
Urinary Anthocyanin Concentration | sampled on day 6, 13, 20, and 27 (participant randomized to different interventions each visit)
  C18 solid-phase extraction (SPE) clean-up methods will be used to isolate anthocyanins and non-anthocyanin low-molecular weight polyphenol metabolites.
Fecal Polyphenol Catabolite Concentration | sampled on day 6, 13, 20, and 27 (participant randomized to different interventions each visit)
  C18 solid-phase extraction (SPE) clean-up methods will be used to isolate anthocyanins and non-anthocyanin low-molecular weight polyphenol metabolites.
Fecal Anthocyanin Concentration | sampled on day 6, 13, 20, and 27 (participant randomized to different interventions each visit)
  C18 solid-phase extraction (SPE) clean-up methods will be used to isolate anthocyanins and non-anthocyanin low-molecular weight polyphenol metabolites.
Urine Creatinine Content | sampled on day 6, 13, 20, and 27 (participant randomized to different interventions each visit)
  The urine creatinine content will be measured by a urinary creatinine colorimetric assay kit (Cayman Chemical).

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Bolling, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT05488886/ICF_000.pdf